CLINICAL TRIAL: NCT05785663
Title: AminoMedixTM for Radiation Kidney Protection During Peptide-Receptor Radionuclide Therapy (PRRT): Phase I, II Clinical Trial
Brief Title: AminoMedixTM for Kidney Protection During Radionuclide Therapy
Status: Completed | Type: Observational
Sponsor: Excel Diagnostics and Nuclear Oncology Center (Other)
Collaborators: Radiomedix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 118766
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Radiation Nephropathy
Keywords: Radiation nephropathy; PRRT; Radiation induced toxicity; 177Lu-DOTATATE; AminoMedix ™

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- I: Subjects received Lysine hydrochloride 26 g ± 5% Arginine hydrochlordie 26 g ± 5% Amifostine trihydrate 0.65 g ± 5%
- II: Subjects received Lysine hydrochloride 39 g ± 5% Arginine hydrochlordie 39 g ± 5% Amifostine trihydrate 0.98 g ± 5%
- III: Subjects received Lysine hydrochloride 52 g ± 5% Arginine hydrochlordie 52 g ± 5% Amifostine trihydrate 1.3 ± 5%
- IV: Subjects received Lysine hydrochloride 60 g ± 5% Arginine hydrochlordie 60 g ± 5% Amifostine trihydrate 1.5 ± 5%

SUMMARY:
This is a phase I, and II, single-center, open-label clinical trial to evaluate the safety and preliminary efficacy information of AminoMedix™ in protecting kidneys from radiation-induced toxicity during Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE in patients with neuroendocrine cancers.

Aims of the study:

1. Evaluation of the safety of AminoMedix ™ infusion.
2. Evaluation of kidney radiation dosimetry with and without AminoMedix™ using 68Ga-DOTATATE PET/CT imaging as a surrogate marker for 177Lu-DOTATATE.
3. Evaluation of the safety and calculation of kidney and tumor radiation dosimetry after AminoMedix™ infusion with low dose 177Lu-DOTATATE in patients with neuroendocrine cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neuroendocrine tumors are eligible to be recruited in this project.
2. Signed informed consent.
3. Patients of either gender, age 18 years or older.
4. Na+, K+, Cl,: within normal range
5. eGFR: > 50 mL/min
6. Serum creatinine: <150μmol/L. Serum creatinine: within normal range or <120μmol/L for patients aged 60 years or older.
7. Negative pregnancy test (urine test or beta-HCG) in women capable of child-bearing.

Exclusion Criteria:

1. Known hypersensitivity to Amifostine, Lysine, Arginine, DOTA, 68Gallium, to DOTATATE or to any of the excipients of 68Ga-DOTATATE.
2. Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 2 days) prior to study imaging. If a patient is on Sandostatin® LAR a wash-out phase of 28 days is required before the injection of the study drug.
3. Pregnant or breast-feeding women.
4. Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
5. Pre-existing cardiovascular or cerebrovascular conditions such as congestive heart failure, ischemic heart disease, arrhythmias, or a history of stroke or transient ischemic attacks.
6. Uncontrolled kidney disease and patients who are under dialysis.
7. Current treatment with potentially nephrotoxic drugs such as aminoglycosides.
8. Less than 24 hours of withdrawal of antihypertensive medications or uncontrolled hypertension, and diabetes at the time of the study.
9. Patients under total or partial parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE in patients with neuroendocrine cancers.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of kidney radiation dosimetry in subjects with and without AminoMedix™ using 68Ga-DOTATATE PET/CT imaging as a surrogate marker for 177Lu-DOTATATE™ | 24 hours to 3 weeks between two dosimetry
  Dosimetry results of 68Ga-DOTATATE in subjects, with and without AminoMedixTM will be compared. Each Subject will be imaged with and without AminoMedixTM 24 hours to 3 weeks apart and the reduction ratio will be calculated

SECONDARY OUTCOMES:
Frequency and Severity of Adverse Events after AminoMedix™ infusion | Subjects will be followed for two weeks following administration of AminoMedix™
  Frequency and severity of treatment-related adverse events as assessed by CTCAE v4.0" in subjects after AminoMedix™ infusion